CLINICAL TRIAL: NCT05840276
Title: Cryoneurolysis Prior to Total Knee Arthroplasty for the Management of Postoperative Pain; A Randomized, Sham-controlled, Trial
Brief Title: Cryoneurolysis Prior to Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cryo_tka
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain; Knee Osteoarthritis; Opioid-Related Disorders
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee; Opioid-Related Disorders | interventions — Cryosurgery; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CRYO (Experimental): Receives cryoneurolysis treatment on the anterior femoral cutanous nerve and the infrapatellar branch of the saphenous nerve.
  Interventions: Device: Cryoneurolysis
- SHAM (Sham Comparator): Receives similar procedures as in CRYO but with no freezing temperatures.
  Interventions: Other: Sham

INTERVENTIONS:
Device: Cryoneurolysis — The VISUAL-ICE uses a combination of argon and helium, to create a highly localized cold zone with temperatures between -20 and -100°C. A probe will be inserted percutaneously at the target AFCN and IBSN guided by ultrasound visualization to accurately determine the location of the nerve and to account for adjacent neurovascular structures and variations in anatomical structures. The target locations are drawn directly on the patients' skin prior to treatment along which a dose of local anesthetic will be injected subcutaneously before treatment. Cryoneurolysis at each target site requires 2 freeze cycles with a duration of 3 mins, and with thaw cycles between 20-40 seconds.
  Other Names: Cryoanalgesia; Cryoneuroablation; Cryoablation
  Arms: CRYO
Other: Sham — A sham needles will be inserted percutaneously at the target AFCN and IBSN guided by ultrasound visualization. The target locations are drawn directly on the patients' skin prior to treatment along which a dose of local anesthetic will be injected subcutaneously before treatment. Sham will simulate cryoneurolysis at each target site for 2 freeze cycles with a duration of 3 mins, and also simulate thaw cycles between 20-40 seconds. No temperature changes will actually occur although the experience and sounds will be similar to cryoneurolysis
  Arms: SHAM

SUMMARY:
Knee osteoarthritis is a major issue worldwide with limited treatment options. Many patients receive knee joint replacement surgery which is considered effective and safe. Nonetheless the period post-surgery is characterized by moderate to severe pain inhibiting early ambulation, motivation and range of motion, compromising rehabilitation, patient satisfaction, and overall outcomes. An optimal strategy of postoperative pain treatment after knee replacement surgery has not yet been established.

Recently, our research center and others have shown that is possible to target the nerves surrounding the knee with a novel treatment called cryoneurolysis. Cryoneurolysis apply low temperatures [-20°C ; -100°C] to a target nerve, which disrupts nerve function and provides potential pain relief. This suggest a potential for cryoneurolysis to significantly improve rehabilitation, reduce opioid intake and overall outcomes after knee replacement surgery.

The primary objective of the current project is to determine the effectiveness of cryoneurolysis in its proposed ability to reduce opioid intake and postoperative pain after knee replacement surgery.

The study is a randomized controlled study with two groups. Group CRYO receives cryoneurolysis prior to knee replacement surgery and group SHAM receives a sham treatment prior to knee replacement surgery. Both groups receive surgery, analgesics and postoperative rehabilitation as per usual.

Efficacy of treatment is evaluated using the change in opioid intake in the CRYO group compared to the SHAM group 14 days after knee replacement surgery. Participants will also be assessed at 90 and 180 days after knee replacement surgery and will include measures on pain, quality of life and function.

DETAILED DESCRIPTION:
INTRODUCTION In Denmark and the rest of Europe, 20% of all chronic pain conditions is related to osteoarthritis (OA) and the incidence of this pathology is likely to increase significantly. The treatment of knee OA typically focuses on pain relief, however the effects of current conservative treatment options remain small to moderate and most are associated with side effects. In many cases patients alternatively may be subjected to partial/total knee arthroplasty (TKA). The number of TKA procedures, in the U.S., is projected to grow by 85% (1.26 million procedures) by 2030. TKA is considered to be an effective treatment for end-stage knee osteoarthritis, however the period post-surgery is characterized by moderate to severe pain. Postoperative pain inhibits early ambulation, motivation and range of motion, compromising rehabilitation, patient satisfaction, and overall outcomes. In this regard, more than 20% of patients have been shown to experience persistent and unchanged pain post-surgery. In an attempt to attenuate postoperative pain, many multimodal approaches have been proposed and implemented, with mixed results however an optimal strategy of postoperative pain treatment after TKA has not yet been established.

Reviewing these results, focus should be on low-risk, minimally invasive pain management. Novel advances in the ability to target the genicular nerves are in that respect promising. Cryoneurolysis has made it possible to apply low temperatures [-20°C ; -100°C] to a target percutaneous peripheral nerve, causing Wallerian degeneration. This disrupts nerve function while structural elements of the nerve bundle remain intact allowing for complete regeneration and functional recovery of the nerve over time. Cryoneurolysis on peripheral nerves has been shown to provide pain relief in a variety of chronic pain conditions such as lumbar facet joint pain, plantar fasciitis, occipital neuralgia, post thoracotomy pain syndrome, and Morton's neuroma.

Recently, our research center and others have shown that is possible to target the superficial genicular nerves with cryoneurolysis and studies have observed a statistically significant reduction in hospital stay, a decrease in prescribed opioids, and less knee symptoms after TKA when cryoneurolysis was provided prior to operation. These results suggest a potential for cryoneurolysis to significantly improve rehabilitation and overall outcomes. Nevertheless, these studies lack adequate power and a control group to confirm its efficacy and safety. In addition, the optimal freezing protocol for cryoneurolysis remains to be outlined. This involves number of cycles, duration, intensity and thaw time which also depends on crucial factors such as nerve target identification, probe placement and anatomical location of the target tissue.

The present study is the first to utilize methodology, that allows for accurate control of the ablation zone in relation to the target genicular nerves. The nerves are identified using electrical nerve stimulation and ultra-sound, which allows for the identification of nerve structures specific for each patient, independent of the inherent variation of neural structures, and also, from a patient security point of view, considers adjacent neurovascular structures and variations in anatomical structures. We have in our center performed 500+ ablations, using the framework, without any serious adverse events.

If cryoneurolysis successfully attenuates postoperative pain, and as a results opioid use, earlier ambulation, improved rehabilitation and overall outcomes - it would have massive socioeconomic implications. Finally, developing and establishing an efficacious and safe protocol for the treatment of pain with cryoneurolysis, is an initial step for its implementation in a much broader context within the field of pain medicine and cryoanalgesia.

OBJECTIVES The primary objective of the current project is to determine the effectiveness of cryoneurolysis in its proposed ability to reduce opioid intake and postoperative pain after TKA.

The secondary objective is to evaluate whether such treatment affects functional performance, quality of life and patient satisfaction.

Finally, development of safe and efficacious freezing protocols for upcoming studies and future research

TRIAL DESIGN This study is a single center, randomized, controlled trial designed to test the efficacy of cryoneurolysis treatment in patients undergoing TKA. The patients will be randomly allocated in either a cryoneurolysis intervention group (CRYO) or a sham group (SHAM) and will be assessed at baseline and after 14 days, 90 days, and 180 days post TKA. The tests will include both patient-reported outcomes (PRO) and objective functional measurements.

Randomization will be performed as computer-generated block randomization with a 1:1 allocation ratio using random block sizes of 2, 4 and 6 in either group CRYO or group SHAM. The randomization restrictions will not be disclosed to ensure allocation concealment and the sequence will be performed by an external co-investigator.

To account for the placebo effect and reduce the risk of bias, the patients, therapists and data-manager will be blinded to the allocation. The allocation code will be concealed in a sealed envelope, that will be available for the surgeon performing the cryoneurolysis procedure only. Blinding will be assured using a sham trial that includes the same procedures as cryoneurolysis treatment but without any freezing temperatures. Thus, visible marks as a result of the procedures in both groups will be similar.

In case of unexpected issues and if deemed absolutely necessary by the investigators and physician, unblinding will occur according to emergency unblinding procedures that will maintain the integrity and confidentiality of the study.

INTERVENTIONS The groups will be allocated to receive either sham or cryoneurolysis treatment. Following intervention and TKA, both the SHAM and CRYO group will receive standard rehabilitation programs, standard analgesics and opioids.

Cryoneurolysis Cryoneurolysis is a minimally invasive procedure and has been in use since the 1960s. The methodology has developed over time, and alongside the advent of ultrasound guided probe insertion, it has become possible to treat multiple chronic pain conditions. The current project involves the novel application and test of cryoneurolysis, in the treatment of OA related pain. The device used to perform the cryoneurolysis treatment is the VISUAL-ICE (Galil Medical, Arden Hills, MN). The rationale behind this device, is based on previous reports showing that low temperature conditions can alter nerve function. This technology allows for reversible destruction of nerves, also known as Wallerian degeneration, that prevents nerve signaling and potentially alleviate pain and motor dysfunction in a number of medical conditions. The severity of nerve damage is dependent on the temperatures used to perform cryoneurolysis. The goal in the current study is the apply temperatures between -20°C to -100°C at which the original structural scaffold of the nerve is preserved, allowing for predictable regrowth of the axon along the epineurium and endoneurium, allowing for the reinnervation of the sensory receptors over time. This regeneration of the nerve is a well-established principle, and means that the nerves' sensory capabilities return.

The VISUAL-ICE uses a combination of argon and helium, to create a highly localized cold zone with temperatures between -20 and -100°C. A probe will be inserted percutaneously at the target AFCN and IBSN guided by ultrasound visualization to accurately determine the location of the nerve and to account for adjacent neurovascular structures and variations in anatomical structures. The target locations are drawn directly on the patients' skin prior to treatment along which a dose of local anesthetic will be injected subcutaneously before treatment. Cryoneurolysis at each target site requires 2 freeze cycles with a duration of 3 mins, and with thaw cycles between 20-40 seconds. A temperature probe will be inserted adjacent to the target nerve and cryoneurolysis-probe to ensure a controlled cooling effect and to control nerve damage.

The sham intervention includes the same procedures as described above but using a sham probe that does not allow for any freezing temperatures.

Total Knee Arthroplasty Primary TKA is performed by trained orthopedic surgeons, using an anterior midline incision and medial parapatellar arthrotomy. Other than cryoneurolysis for CRYO group, all patients received similar perioperative pain management.

Rehabilitation All patients will be subjected to a standard rehabilitation protocol. On the operation day the patients begin to be mobilized with the help of the physiotherapists and the nursing staff and are instructed in standard exercises. All patients receive the exercise plan in written form. If needed, the patients receive more intensive rehabilitation during the stay and/or have a longer stay. After the discharge from the hospital, all patients are invited to a two-week and a three-month control with a physiotherapist.

Analgesics and opioids During TKA all patients receive a standard protocol of local infiltrative anesthesia (LIA) with 150ml 2mg/ml Ropivacain with Adrenalin: 50 ml in the posterior capsule before the cementing, 25 ml in the medial ligaments, 25 ml in the lateral ligaments and 50 ml in subcutis during the skin closure.

After the operation, all eligible patients receive standard protocol pain medication: Paracetamol 1000 mg x 4, Ibuprofen 400 mg x 4, Morphine 10 mg if necessary, max. 80 mg per day. Patients who reach maximal dose of Morphine tablets begin to receive depot from the next day.

DATA COLLECTION METHODS Intake of analgesic medicine Opioid intake will be evaluated during the first 14 days after knee arthroplasty and will be assessed using a patient medicine intake questionnaire. Further use and prescriptions will be controlled via national recorded medical records (Fælles Medicin Kort) of prescribed medicine during the project period. Patients receive a standard analgesic prescription post TKA comprising ibuprofen, paracetamol, morphine and, if needed, depot morphine.

Pain Pain intensity will be assessed using the VAS pain intensity score. VAS is a research and clinical tool widely used in diverse populations33. VAS consists of a continuous scale, typically 100 mm in length, anchored by two verbal descriptors, "no pain" for the score of zero and "worst pain imaginable" for the score of 100. VAS is a self-reported tool where the respondent is asked to mark the point representing their current pain intensity. This provides a score (the distance between 0 and the respondents mark) in the range [0-100mm], which takes <1 minute to complete, requires little training to administer and score and has been reported to be reliable34. In addition to intensity, other pain characteristics such as location, duration and type will be recorded as well.

Functional performance Functional performance will be evaluated by the 30 second chair-stand test, the 40m fast-paced walk test, the 9-step stair-climb test and MVC force. The 30 second chair-stand test consists of repeated sit-to-stand movement for a duration of 30 s. The starting position is seated, with feet placed flat on the floor, shoulder width apart and with the arms crossed on the chest. The position change to standing, with hips and knees fully extended, followed by sitting back down, with bottom fully touching the seat. The test is performed with usual footwear and the chair should be with a straight back, with no arms, seat height 43 cm, placed against a wall. In cases where the movement cannot be performed even once, the hands are allowed to be placed on the legs or a regular mobility aid can be used - the result is then reported as an adapted test score. The outcome is the total number of complete chair stands performed for the duration of the task (one chair stand represents a stand followed by a sit movement).

The 40m fast paced walk test consists of walking as fast as possible, but still safely, along a 10 m marked walkway, then turning around a cone / tape and return. This is then repeated for a total distance of 40 m. The test is performed with usual footwear and regular walking aid is allowed and recorded. The outcome is expressed as speed. i.e. walking distance (40m) divided by the time to perform the task (s). Timing is paused during turns.

The 9-step stair-climb test consists of the ascend and descend a flight of stairs as fast as possible, but still safely. The flight of stairs preferably has 9 steps, step height appx. 20 cm, with hand rails. The test is performed with usual footwear and regular walking aid is allowed and recorded. The outcome is the total time to perform the task (s).

Quadriceps strength will be assessed measuring isometric MVC force of the knee extensors. Patients will be seated in a chair with knee and hip flexed at 90° and with the pelvis and chest restrained by straps. A non-extensile chain attached to the back of the chair and connected to a force transducer will be placed just proximal to the malleolus. The patient will then be asked to perform three knee extensions pushing as hard as possible against the chain, with 1 min rest in between. The highest peak value out of the three MVCs will be taken as the MVC force.

PRO-data PRO-data will be recorded using the Oxford Knee Score (OKS) developed and validated specifically to asses pain and function after knee arthroplasty. The OKS consists of 12 questions about the patients' level of function, activities of daily living and pain over the preceding four weeks.

Health-related quality of life will be assessed using the SF-36 questionnaire. The SF-36 includes eight dimensions; physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. It's a validated and widely used questionnaire.

Pain catastrophizing will be assessed using the pain catastrophizing scale. Questions indicate thoughts and feelings when experiencing pain and also includes subscales on rumination, magnification and helplessness.

Adverse effects All adverse effects will be recorded using both prespecified symptom inventories and open-ended questions on both cryoneurolysis and morphine intake.

STATISTICAL METHODS To evaluate the empirical distributions of the continuous outcomes, visual inspection of the studentized residuals will be applied to evaluate whether the assumption of normality is reasonable.

The treatment groups will be examined for comparability based on baseline demographic and prognostic measures. An Intention-To-Treat (ITT) analysis will be used for all allocated patients and a mixed effects model will be used on the continuous outcome measures to determine the effects of cryoneurolysis treatment from baseline to post treatment and follow-ups [Between groups factor: CRYO vs SHAM, within groups factor: time]. The model will use robust estimation methods to account for outliers. All P-values < 0.05 will be considered statistically significant.

HARMS Any adverse effects will be recorded and reported according to the guidelines of the Regional Committee on Health Research Ethics for Southern Denmark within 7 days. Once a year the investigator will report all expected and unexpected adverse effects that have occurred during that period, with an evaluation of patient safety.

Cryoneurolysis Cryoneurolysis is a minimally invasive procedure that cause Wallerian degeneration where the nerve structure and conduction are disrupted while structural elements of the nerve bundle remain intact by applying temperatures between -20°C to -100°C. This temperature range results in reversible destruction of the nerves that allow for complete regeneration and functional recovery. In a preclinical study, Hsu and Stevenson 39 examined the nerves in rats histologically post cryoneurolysis treatment and observed significant axonal regeneration and remyelination after 8 weeks and complete axonal regeneration 16 weeks post cryoneurolysis as compared to baseline. Thus, the target nerves suffer no permanent damage in rats. The regeneration of sensory peripheral nerves after damage is a well-established principle but depends on the nature of the nerve damage. Regeneration predominantly depends on the integrity of the surrounding endoneurial, perineurial and epineurial structures, which has been shown to be unaffected in animal models at the temperature range -20°C to -100°. This is likely explained by a remarkable resilience of collagen and fibroblasts to hypothermia. In contrast to other therapies such as ablation with heat, cryoneurolysis induces a mild lesion. No studies have investigated the histological results of cryoneurolysis in humans, however studies investigating human clinical results concurrently with animal models suggests that the effect of cryoneurolysis is comparable. This also means that pain sensation might return over time and studies do show a gradual increase in sensory capabilities after cryoneurolysis treatment. Cryoneurolysis is not a curative to chronic pain. The current study will insert a temperature probe, using ultra-sound, adjacent to the target nerve and cryoneurolysis-probe to ensure a controlled cooling effect, at the specified temperatures, to control nerve damage and increase safety. In addition, the nerves of interest (IBSN, AFCN) is located on the opposite side of the knee than the proprioceptive nerves surrounding the knee. Proprioception will therefore not be affected.

Adverse effects associated with cryoneurolysis treatment include frostbite to skin, alopecia, depigmentation of skin, and damage to surrounding structures. These effects are often mild and can be avoided with careful technique during the procedure, with prober thaw options and meticulous skin precautions. The procedure in the current study will be performed by a trained orthopedic surgeon. Because cryoneurolysis is an invasive procedure (however minimal), adverse effects also include bleeding, bruising, redness, infection and development of an insensate area at the site of treatment. A recent study investigating cryoneurolysis in knee OA (n=180), observed side effects such as altered sensation (20%), crusting (5%), itching (5%), local pain (21%), numbness (53%), swelling (36%), tenderness on palpation (17.8%) and tingling (11%), in addition to the aforementioned. The majority of these effects were categorized as mild in severity and were resolved within 30 days. Another study reported no complaints of persistent numbness or other neurologic effect at the three-months follow-up.

The current project will use ultrasound visualization to accurately determine the location of the nerve and to account for adjacent neurovascular structures and variations in anatomical structures.

There is a risk for neuroma formation or neuritis, however these are very rare. Two different reviews stated that there has been no reported cases of permanent nerve damage as a result of cryoneurolysis and so far there is only one reported case of neuritis after cryoneurolysis treatment47. This is in line with what the authors of the current clinical protocol have observed in their search through the literature. The investigators in the present study have extensive experience providing treatment with cryoneurolysis having performed 500+ ablations, as part of a similar and previously approved protocol (S-20180089) and have not reported any serious adverse events.

Analgesics and opioids Opioids are widely used to attenuate both moderate and severe pain. Nevertheless these have important limitations that should be taken into account. Opioid-related adverse effects include but are not limited to, opioid use disorder, nausea, constipation, dry mouth, dizziness, drowsiness, falls, lack of energy, postoperative infection, endocrinopathy, altered immune function, respiratory depression, misuse, abuse.

RESARCH ETHICS The project will be conducted according to the declaration of Helsinki. Furthermore, the project will be registered in ClinicalTrials.gov.

Given the study design, eligibility criteria and safety measures, the current project does not include special risks for the participating patients. The majority of risks does not require medical attention and serious adverse effects as a result of local anesthetics and cryoneurolysis are very rare. A clinical expert will be available to respond to any enquiries or adverse effects. If adverse effects are identified, patients will be referred to the relevant clinical department and care will be provided as needed as part of the Danish health security system. The project is covered in accordance with Danish Patient Compensation Act. . The investigators will review the trial processes and data continuously.

The potential benefits of the current project include increased functional capacity and quality of life as a result of significant pain relief, reduced opioid intake and improved rehabilitation. This could have a significant impact on patients' lives as well as significant socioeconomic consequences.

The inclusion of a sham group is necessary to test the hypothesis because of the large reported placebo effects in OA trials51. In addition, the associated risks are minimal and the nature of misleading, in regards to the administration of the sham trial, will be adequately disclosed and accepted by the patient during the informed consent process. The sham group is implemented according to current standards

PROTOCOL AMENDMENTS To maintain trial integrity, changes to the protocol that might impact the conduct of the study, including changes of study objectives, design, patient population, sample size or other relevant procedures will be formally reported to the Regional Committee on Health Research Ethics for Southern Denmark and trial registries.

DATA MANAGEMENT All data will be kept electronically and filed according to a participant code. Data entry will always be handled by the same investigator, who will use unambiguous and standard terminology based on predefined study forms. Complete back-up of all data will be performed regularly and stored on secured servers in the Region of Southern Denmark via encrypted connection and restricted access that fulfil the demands for data security. Data will be stored for a duration of 10 years.

CONFIDENTIALITY All information related to the study, including patient information, will be stored securely, with restricted access, at the Hospital of South West Jutland, University hospital of Southern Denmark, Esbjerg, Denmark. The data will be identified by a coded identity number to maintain participant confidentiality and stored separately. The investigators are under duty of confidentiality.

The project will be reported to the Danish Data Protection Agency and will be handled according to the General Data Protection Regulation (GDPR) and the Danish Data Protection Act.

ACCESS TO DATA The full data set will be available on request to the lead investigators. All shared data will be fully anonymized.

ECONOMY The current project was initiated by Carsten Kock-Jensen, MD, CRPS Center South, Hospital of South West Justland and is funded by Boston Scientific. Funds are paid to a specific research account administered by the Hospital of South West Jutland, University hospital of Southern Denmark, Esbjerg, Denmark, and is subject to public audit under Rigsrevisionen.

The current project is independent of the grants listed and there are no conflicts of interests.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral, primary total knee arthroplasty
* Age ≥ 18y
* Written and oral understanding of Danish.

Exclusion Criteria:

* Contraindications against ibuprofen or paracetamol, for example previous gastric ulcer, or known renal failure (eGRF < 60 ml/kg/1,73m2), known thrombocytopenia (< 100 bil/l); or against treatment with morphine
* History of neuropathic pain
* Previous recipient of cryoneurolysis for the knee
* Patients with daily use of high dose opioid (> oral morphine 30 mg/day or oxycodone 30 mg/day or tramadol 150 mg/day) or any use of other opioids including methadone and transdermal opioids
* Uncontrolled serious disease (cancer, diabetes, etc.)
* Disease associated with reactions to cold, such as cryoglobulinemia, cold urticarial and Reynaud's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Opioids | 14 days after total knee arthroplasty
  Oral morphine intake after total knee arthroplasty in CRYO compared to SHAM

SECONDARY OUTCOMES:
Pain scores on the visual analogue scale | 14, 90 and 180 days after total knee arthroplasty
  Pain score measured on the visual analogue scale after total knee arthroplasty in CRYO compared to SHAM. The visual analogue scale is anchored from 0 (no pain) to 10 (worst pain imaginable)
Adverse effects | 14, 90 and 180 days after total knee arthroplasty
  Adverse effects from cryoneurolysis in CRYO compared to SHAM
Opioid-related adverse effects | 14, 90 and 180 days after total knee arthroplasty
  Opioid-related adverse effects in CRYO compared to SHAM
Pain and Function | 90 and 180 days after total knee arthroplasty
  Patient-reported outcome on pain and function using Knee Oxford Score
Quality of Life using SF-36 | 90 and 180 days after total knee arthroplasty
  Patient-reported outcome on quality of life using SF-36
Pain catastrophizing | 90 and 180 days after total knee arthroplasty
  Patient-reported outcome on pain catastrophizing using the questionnaire: pain catastrophizing scale
Function, Chair-stand test | 90 and 180 days after total knee arthroplasty
  Repeated sit-to-stand movement for a duration of 30 s.
Function, walk test | 90 and 180 days after total knee arthroplasty
  walking as fast as possible, but still safely, along a 10 m marked walkway, then turning around a cone / tape and return for a total distance of 40 m.
Function, Stair test | 90 and 180 days after total knee arthroplasty
  The ascend and descend a flight of stairs as fast as possible, but still safely

CONTACTS AND LOCATIONS:
Overall Officials: Niels-Peter B Nygaard, PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark; Carsten Kock-Jensen, MD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of Southwest Jutland, Esbjerg, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The full data set will be available on request to the lead investigators. All shared data will be fully anonymized.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after completion and publication of the study results.
Access Criteria: Data must adhere to the Danish Data Protection Agency and must be handled according to the General Data Protection Regulation (GDPR) and the Danish Data Protection Act.